CLINICAL TRIAL: NCT05277584
Title: Prediction of Timely Evolution of Plasma Sodium in Treatment of Hyponatremia - Post Hoc-analysis of the Hyponatremia Registry
Brief Title: Analysis of Factors Determining Increase of Serum Sodium in Hyponatremic Patients
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: Department of Mathematics and Computer Science, University of Technology Eindhoven (Unknown)
Responsible Party: Principal Investigator, Volker Burst, Prof. MD, University of Cologne
Other Study IDs: 01
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Hyponatremia
Keywords: Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hyponatremia

SUMMARY:
The aim of this study is to further analyse the dataset of the Hyponatremia Registry, a multicenter, prospective, observational study conducted between September 2020 and February 2013 in the United States of America and the European Union. The primary interest was to provide evidence to investigators' hypothesis that baseline sodium levels are a predominant factor determining the rapidity of sodium increase irrespective of the given treatment. Further investigators aimed to identify other independent predictors of the increase of plasma sodium upon treatment.

DETAILED DESCRIPTION:
Hyponatremia is the most common electrolyte disorder in outpatients and hospitalized patients. Overly rapid sodium increase is associated with increased risk for osmotic demyelination. Smaller analyses have suggested that the slope of the sodium increment is higher with lower baseline sodium levels but this has not been confirmed in large datasets. Investigators have recently published the results of analysis on patients from the Otsuka HN-Registry on thiazide-induced hyponatremia (cooperation with Otsuka). In that dataset was founded the same association and there had been hints that this relationship holds true for all kinds of treatment including no treatment at all.

Investigators took the datasets of those patients presenting with Hyponatremia that could be classified into one etiology group by the treating physician for further analysis. Patients with euvolemic, hypervolemic, hypovolemic or thiazide-associated HN were included in investigators' analysis. Furthermore investigators only considered those cases in which the patient record provided at least one documented plasma [Na+] within <25 hours after the first plasma [Na+] ≤130mEq/L had been measured.

All variables collected in the HN registry were included in the data base. All available information on ingested or administered solutes was recorded. Linear mixed effects models were applied to conduct multivariable repeated measures analyses.

Following questions are to be answered in this study

1. Is the baseline sodium level a predominant factor determining the rapidity of sodium increase?
2. Ist he rapidity of sodium increase correlated to the given treatment?
3. Can other predominant factors of slope of sodium increase be determined?

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypotonic hyponatremia <130 mmol/l enrolled in the Hyponatremia Registry and classified as Euvolemic Hyponatremia, Hypervolemic Hyponatremia, Hypovolemic Hyponatremia or Thiazide associated Hyponatremia-Group

Exclusion Criteria:

* Patients, who could not be assigned to one etiology group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypotonic hyponatremia <130 mmol/l enrolled in the Hyponatremia Registry (NH-Registry)
Sampling Method: Probability Sample
Enrollment: 3460 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Predictors of [Na+] slope due to therapy | Enrollment
  Assessing Evolution of plasma sodium within the first 24 hours after commencement of therapy to determine predictors for velocity of [Na+] increase.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — Department II of Internal Medicine, University of Cologne
Locations (1):
- Department II of Internal Medicine,University of Cologne, Cologne, Germany